CLINICAL TRIAL: NCT05496387
Title: Effect of Neuromobılızatıon on Stiffness of Scıatıc Nerve in Patients With Nonspecific Low Back Pain: Randomized Controlled Trial
Brief Title: Effect of Neuromobılızatıon on Stiffness of Scıatıc Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yunus Emre Tutuneken, Lecturer, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Neuromobılızatıon; Stiffness; Scıatıc Nerve; Nonspecific Low Back Pain

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled, double-blinded study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator did not collect pre-and post- neuromobilization techniques data and the patients were not aware of whether they had been allocated to tension or sliding group. Participants' evaluation and interventions were performed by different investigator. Participants were trained at different places.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Group One (Experimental): Sciatic nerve neuromobilization techniques (tension) was applied to the dominant side lower extremities of all participants in the study.
  Interventions: Other: Sciatic nerve neuromobilization techniques
- Study Group Two (Experimental): Sciatic nerve neuromobilization techniques (sliding) was applied to the dominant side lower extremities of all participants in the study.
  Interventions: Other: Sciatic nerve neuromobilization techniques
- Control Group (Sham Comparator): No application was applied to the sham group
  Interventions: Other: Sciatic nerve neuromobilization techniques

INTERVENTIONS:
Other: Sciatic nerve neuromobilization techniques — Sciatic nerve neuromobilization techniques (tension and sliding) was applied to the dominant side lower extremities of all participants in the study. While the participant was trying to bring her chin closer to her chest by flexing her head and neck, she simultaneously brought her foot to dorsiflexion. After waiting 30 seconds in this tense position, the ankle, head and neck returned to neutral position and relaxed. 3 sets were repeated with 1 minute rest breaks. Sciatic nerve sliding was applied in the same starting position as tension. While the participants was trying to bring her chin closer to her chest by flexing her head and neck, she simultaneously brought her foot to plantar flexion.

SUMMARY:
Low back pain (LBP) is a common symptom that can be a health problem in worldwide. Studies have shown that 70% to 80% of all people are affected at least once in their lives. Although it is common, the cause of the pain has often not been determined and is referred to as non-specific LBP. The lumbar range of motion decreases, trunk flexion is limited, postural control and muscular stiffness are affected in individuals with LBP. Recent studies have shown that people with LBP have altered nerve properties in the sciatic nerve. It was observed that the cross-sectional area of the sciatic nerve decreased and its stiffness increased.

Peripheral nerve tissues are faced with great tension and compressive forces that occur in daily life activities and sports activities. To maintain the normal function of the nervous system, it must have the ability to resistance to tension, easy to slide in the environment it is in and withstand compressive forces. In case of not being able to resist the pressure exerted by surrounding tissues such as bone, tendon, muscle, fascia, there may be distortions in the shapes of neural structures.

Neuromobilization, one of the manual therapy techniques, is used in impingement syndromes of peripheral nerves and neuropathies. Neuromobilization aims to regain the normal mechanical properties of the nerve by using limb movements, motion and position of the joint. There are two methods of neuromobilization techniques; sliding and tension. Sliding involves combinations of movements that lengthen the nerve bed in one joint and reduce the length of the nerve bed in the next joint, while tension is done by stretching both ends of the nerve bed. Neuromobilization structures the balance between the relative movements of the neural tissues and the surrounding mechanical interface, allows the reduction of internal pressure in the neural tissue, and thus optimum physiological functions are regulated. The mechanism of action of neuromobilization is thought to be to increase intraneural circulation, improve axoplasmic flow and connective tissue viscoelasticity, and reduce hypersensitive areas.

Neuromobilization techniques are extensively used in clinical settings during the therapy of patients with sciatica, with favorable effects on pain and impairment. However, the mechanical implications of neuromobilization in human nerves are poorly understood. Two investigations that used SWE to measure sciatic nerve stiffness in healthy adults following prolonged slump positions came up with conflicting conclusions. It has been determined that there are different opinions on the effects of slump neuromobilizations in sciatic nerves. Considering that slump neuromobilization techniques are frequently used for therapeutic, it should be appropriate to determine their effects on the sciatic nerve.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of nonspecific LBP Having pain for at least 3 months

Exclusion Criteria:

Obesity Pregnancy Specific disorders of the lumbar spine such as disc problems Spinal stenosis Having indication for surgery Any recent or old significant trauma of the lumbar region Any systemic inflammatory disease Having neurological problems Any forms of physiotherapy within 6 months before the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
SWE Imaging | 4 week
  Longitudinal ultrasound SWE images of the sciatic nerve will be taken bilaterally with a linear array probe in the prone position. By selecting the largest area within the epineurium boundaries in the elastographic window, a rapid area of interest will be determined on the sciatic nerve in each clip. This approximation will be made for each frame to ensure that the area of interest is not affected by nerve movement throughout the maneuvers. The color pixels of each elastogram will be converted to SWV values using the appropriate scale (maximum 17.0 m/s) (15).

SECONDARY OUTCOMES:
The Sit-and-Reach Test | 4 week
  Flexibility of the back and legs will be assessed using the sit and lie down test. A specially designed box will be used for the test. The participant will sit in front of the 23 cm box with their knees bent and their legs together. The person has extended his arm as far as he can and will hold it there for two seconds.
The Straight Leg Raise (SLR) Test | 4 week
  During the test, the participants will be placed in the supine position with their knees in full extension and the other knees in half flexion. He will be asked to try to stretch his hip by raising his leg up. The test will be terminated at the point where he feels pain and tension in the waist and hip.
The Vertical Jump Test | 4 week
  During the counter move, participants stand with their feet shoulder-width apart, with equal weight distribution on both feet, and will make a mark at the highest point they can reach. Participants will then mark the highest point they can reach by jumping by bending their knees and ankles. The distance between these two marks will be measured in centimeters and recorded.
The 3-Step Forward Test | 4 week
  Participants will prepare by bending one knee just behind the starting line and lifting the leg off the ground. Participants performed three jumping moves: jumping on the starting leg, stepping on the other leg, and a double jump. The distance between the starting line and the heel of the foot closest to the line was measured and will be recorded in centimeters.
The Flamingo Balance Test | 4 week
  Participants will stand on the beam, balancing on one leg with bare feet; the other leg is flexed at the knee and the foot is kept close to the hip and the hands will be held on the pelvis. After a trial period of 1 minute, the person will do 3 trials with eyes open on both legs.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided